CLINICAL TRIAL: NCT02252926
Title: Clinical Trial With Lozenges as Local Anesthetic Treatment for Head/Neck Cancer Patients With Oral Mucositis
Brief Title: Local Anesthetic Treatment of Oral Pain in Patients With Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Moberg Pharma, Sweden (Unknown)
Responsible Party: Principal Investigator, Claus Andrup Kristensen, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P2HNC01
Record Dates: First submitted 2014-09-10; First posted 2014-09-30 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Mucositis
Keywords: Anesthetics, Local; Bupivacaine; Lozenge; Administration, Topical
MeSH Terms: conditions — Mucositis | interventions — Bupivacaine; Morphine; Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine lozenge (Active Comparator): The patients can take up to eight 25 mg bupivacaine lozenges (max. every second hour in the awake hours) a day for seven days. The patients can use concomitant systemic pain treatment (e.g. morphine).
  Interventions: Drug: Bupivacaine
- Standard treatment (Other): The patients will be treated with the currently used standard pain treatment (lidocaine viscous solution, morphine, paracetamol, NSAID, gabapentin). The anesthetics are being administered at the physician's discretion.
  Interventions: Drug: Standard treatment (lidocaine viscous solution, morphine, paracetamol, NSAID, gabapentin)

INTERVENTIONS:
Drug: Bupivacaine — 25 mg bupivacaine lozenge
  Arms: Bupivacaine lozenge
Drug: Standard treatment (lidocaine viscous solution, morphine, paracetamol, NSAID, gabapentin) — Standard treatment includes lidocaine viscous solution, morphine, paracetamol, NSAID, gabapentin
  Arms: Standard treatment

SUMMARY:
Oral mucositis is a damage to the mucosa of the oral cavity and pharynx. It is a serious and painful adverse effect caused by the radio therapy and/or chemo therapy patients with head and neck cancer receive. The pain caused by oral mucositis can be difficult to treat as the current treatment with opioids is not sufficient and can cause adverse effects.

Our hypothesis is that treatment with a local anesthetic lozenge with bupivacaine can reduce the oral pain caused by mucositis compared with the current standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with head/neck cancer and starting radio therapy treatment
* age between 18 and 80 years (both included)
* able to talk, read and understand Danish
* ability to give informed consent

Exclusion Criteria:

* known hypersensitivity towards bupivacaine or other local anesthetics of the amide type
* pregnancy
* women breastfeeding a child

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction of oral and pharyngeal pain measured on Visual Analogue Scale (VAS) | 7 days
  The primary outcome measure is the mean VAS score for the patients in the bupivacaine lozenge group compared with the mean VAS score for the patients in the standard treatment group.
  The lozenge group measures VAS before and 60 min. after administration of a lozenge for seven days. The standard treatment group measures VAS every second hour for seven days.

SECONDARY OUTCOMES:
Duration of the effect of the lozenge | 7 days
  Mean value of the pain score (VAS) measured 120 minuts after the administration of a lozenge for the patients receiving the lozenges compared with the mean value of the pain score (VAS) measured every second hour for the patients receiving the standard treatment.
Effect of the bupivacaine lozenge | 7 days
  The difference in pain score (VAS) between the first score in the morning before the first lozenge of the day and the score 60 minuts after the administration of the lozenge. Pain is scored both in the oral cavity and the pharynx.
Safety: Peak plasma concentrations of bupivacaine | 90 minutes
  The first ten patients receiving the bupivacaine lozenge will on day seven (the last day of their treatment period) get blood samples drawn before a lozenge is administrated and at time 30 min, 60 min. and 90 min. after the administration.

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Kristensen, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Jens Bentzen, MD, Principal Investigator — Department of Oncology Herlev Hospital, Denmark
Locations (2):
- Denmark (2):
  - Department of Oncology, Rigshospitalet, Copenhagen
  - Department of Oncology, Herlev Hospital, Denmark, Herlev

REFERENCES:
- [Derived] Mogensen S, Treldal C, Kristensen CA, Bentzen J, Lawson-Smith L, Petersen J, Andersen O. Effect of bupivacaine lozenges on oral mucositis pain: a randomized controlled multicenter phase II study. Pain Rep. 2017 Aug 23;2(5):e619. doi: 10.1097/PR9.0000000000000619. eCollection 2017 Sep. PMID 29392234